CLINICAL TRIAL: NCT02530970
Title: A Post Market Observational Study to Obtain Additional Information on the Use of Cormatrix® Cangaroo ECM® Envelope
Brief Title: A Post Market Study on the Use of Cormatrix® Cangaroo ECM® (Extracellular Matrix) Envelope
Acronym: SECURE
Status: Completed | Type: Observational
Sponsor: Elutia Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-PR-1110
Record Dates: First submitted 2015-08-18; First posted 2015-08-21 (Estimated); Results first posted 2020-03-11 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of the SECURE Study is to actively gather additional information on the use of the CorMatrix® CanGaroo ECM® Envelope in a post market observational study.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have received CorMatrix® CanGaroo ECM® Envelope for an implantable electronic device placement.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects who have received CorMatrix® CanGaroo ECM® Envelope for an implantable electronic device placement.
Sampling Method: Non-Probability Sample
Enrollment: 1025 (Actual)
Dates: Start 2015-10; Primary Completion 2017-12 (Actual); Study Completion 2018-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Green, Study Director — Corvivo Cardiovascular, Inc.
Locations (39):
- United States (39):
  - Advanced Cardiovascular, LLC, Alexander City, Alabama
  - Heart & Rhythm Solution, Chandler, Arizona
  - Cardiac Electrophysiology/St. Joseph, Phoenix, Arizona
  - Arizona Heart Rhythm Center, Phoenix, Arizona
  - Little Rock VA Clinic, Little Rock, Arkansas
  - Mercy Heart & Vascular, Rogers, Arkansas
  - Stockton Medical Center, Stockton, California
  - St. Joseph Heritage Medical Group, Tustin, California
  - Bay Pines VA, Bay Pines, Florida
  - Bethesda, Delray Beach, Florida
  - Florida Heart & Rhythm Specialists, Fort Lauderdale, Florida
  - Baptist Heart Specialists, Jacksonville, Florida
  - UF Health Jacksonville, Jacksonville, Florida
  - Cardiovascular Institute of NW Florida, Panama City, Florida
  - Baptist Healthcare Cardiology, Pensacola, Florida
  - Cardiology Associates, Albany, Georgia
  - Athens Cardiology Group, Athens, Georgia
  - North Georgia Heart Foundation, Gainesville, Georgia
  - Georgia Arrhythmia Consultants, Macon, Georgia
  - The Queen's Medical Center, Honolulu, Hawaii
  - Central DuPage Hospital, Winfield, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Wayne State University Physician Group, Detroit, Michigan
  - St. John Providence, Detroit, Michigan
  - Cardiology Institute of Michigan, Flint, Michigan
  - Advanced Cardiovascular Clinic, Flushing, Michigan
  - Sparrow Thoracic Cardiovascular Institute, Lansing, Michigan
  - HeartPlus Center, Jackson, Mississippi
  - Sanger Heart & Vascular, Concord, North Carolina
  - Carolina East Heart Center, New Bern, North Carolina
  - NC Heart & Vascular, Raleigh, North Carolina
  - Novant Health Winston-Salem Cardiology, Winston-Salem, North Carolina
  - University of Oregon Health Science Center, Portland, Oregon
  - Wellspan Heart & Vascular, York, Pennsylvania
  - AnMed Health Arrhythmia Specialists, Anderson, South Carolina
  - South Carolina Heart Center, Columbia, South Carolina
  - Carolina Heart Specialists, Lancaster, South Carolina
  - Carolina Cardiology Clinical Research, Rock Hill, South Carolina
  - UT Health Science Center - EP Heart, The Woodlands, Texas

REFERENCES:
- [Derived] Deering TF, Catanzaro JN, Woodard DA. Physician antibiotic hydration preferences for biologic antibacterial envelopes during cardiac implantable device procedures. Front Cardiovasc Med. 2022 Dec 22;9:1006091. doi: 10.3389/fcvm.2022.1006091. eCollection 2022. PMID 36620632

RESULTS

PARTICIPANT FLOW:
Groups:
- CanGaroo: Data collection for information on the use of CorMatrix CanGaroo ECM Envelope
Period: Overall Study
Arm/Group | CanGaroo
Started | 1025
Completed | 891
Not Completed | 134
Not completed — Adverse Event | 8
Not completed — Lost to Follow-up | 88
Not completed — Physician Decision | 5
Not completed — Withdrawal by Subject | 14
Not completed — Death | 6
Not completed — Hospitalization | 1
Not completed — Insurance | 2
Not completed — Explant | 2
Not completed — Change in Provider | 5
Not completed — Relocation | 3

BASELINE CHARACTERISTICS:
Arm/Group | CanGaroo
Number analyzed (Participants) | 1025
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 257
  >=65 years | 768
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.9 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 392
  Male | 633
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32
  Not Hispanic or Latino | 990
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7
  Asian | 17
  Native Hawaiian or Other Pacific Islander | 8
  Black or African American | 175
  White | 797
  More than one race | 2
  Unknown or Not Reported | 19
Region of Enrollment [Number; unit: participants]
  United States | 1025
Risk Factors for Infection [Count of Participants; unit: Participants]
  None | 103
  Systemic Anticoagulants | 233
  Chronic Steroid Use | 14
  Renal Insufficiency | 115
  Diabetes | 301
  Prior Device Infection | 18
  Peripheral Vascular Disease | 80
  Pocket Re-entry | 5
  Obesity | 387
  Malnutrition | 12
  Smoker | 121
  Congestive Heart Failure | 450
  Malignancy | 42
  3 or More Leads | 28
  2 or More Risk Factors | 678
  Other | 180
  Temporary Pacing | 68
  Device Replacement/Revision | 377
IV Antibiotic Used Prior to Procedure [Count of Participants; unit: Participants]
  Yes | 938
  Unknown | 50
  No | 37
Pre-Procedure Temporary Pacing [Count of Participants; unit: Participants]
  No | 823
  Unknown | 134
  Yes | 68
Surgical Glue Used in Procedure [Count of Participants; unit: Participants]
  No | 677
  Yes | 321
  Unknown | 27
Procedure Types [Count of Participants; unit: Participants]
  De Novo Pacemaker | 324
  De Novo ICD | 158
  De Novo CRT-P | 27
  De Novo CRT-D | 93
  Pacemaker Replacement | 122
  ICD Replacement | 71
  CRT-P Replacement | 4
  CRT-D Replacement | 71
  Upgrade Pacemaker to ICD | 13
  Upgrade Pacemaker to CRT-P | 21
  Upgrade Pacemaker to CRT-D | 27
  Upgrade ICD to CRT-D | 47
  Downgrad CRT-D to ICD | 1
  Lead Revision/Replacement Only | 36
  Pocket Revision Only | 10

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With ECM Related Adverse Events
Description: ECM related adverse events were collected at all study visits.
Time Frame: Participants were followed for an average of 235.0 days.
Population: Analysis population includes all study participants.
Measure: Count of Participants; unit: Participants
Groups:
- CanGaroo: Arm/group includes all study participants.
Arm/Group | CanGaroo
Number analyzed (Participants) | 1025
Participants
  Possibly Related to CanGaroo | 14
  Probably Related to CanGaroo | 2

2. Primary Outcome: Number of Participants With Major Pocket Infections
Description: Incidence of major pocket infection included those with cellulitis in the region of the CIED pocket with wound dehiscence, erosion or purulent drainage, 2) deep incisional or organ/space (pocket) surgical site infection, 3) persistent bacteremia or 4) endocarditis.
Time Frame: Participants were followed for an average of 235.0 days.
Population: Analysis population includes all study participants.
Measure: Count of Participants; unit: Participants
Arm/Group | CanGaroo
Number analyzed (Participants) | 1025
Participants | 12

ADVERSE EVENTS:
Time Frame: Participants will be followed for an expected average of 3 months
Arm/Group | CanGaroo
All-Cause Mortality (participants affected / at risk) | 17/1025
Serious Adverse Events (participants affected / at risk) | 40/1025
Other Adverse Events (participants affected / at risk) | 0/1025
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CanGaroo (N=1025)
Pain (General disorders) | 5 (5)
Heart Failure (Cardiac disorders) | 1 (1)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Cardiac disorders) | 2 (2)
Superficial Cellulitis (Skin and subcutaneous tissue disorders) | 2 (2)
Pocket Erosion (Surgical and medical procedures) | 1 (1)
Pocket Infection (Infections and infestations) | 12 (12)
Hematoma (Vascular disorders) | 5 (6)
Urinary Tract Infection (Renal and urinary disorders) | 1 (1)
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Lead Issues (Surgical and medical procedures) | 1 (1)
Inappropriate ICD Shocks (Surgical and medical procedures) | 1 (1)
Palpitations & Shortness of Breath (Cardiac disorders) | 1 (1)
Congestive Heart Failure/Renal Failure (Cardiac disorders) | 1 (1)
Superficial CIED Infection (Infections and infestations) | 2 (2)
Suicidal Ideation (Psychiatric disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
NSTEMI (Cardiac disorders) | 1 (1)
Seroma (Cardiac disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
It was single-arm study thereby precluding the possibility of direct comparisons with a control. Also, a longer follow-up would allow for the confirmation of the long-term efficacy of the CanGaroo envelope.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/70/NCT02530970/Prot_SAP_000.pdf